CLINICAL TRIAL: NCT03197805
Title: Prospective Study Assessing the Impact of RNA Genomic Profile Defined by a Genomic Test on Treatment Decision-making in Breast Cancer Patients With an ISH Equivocal HER2 Status- EQUIVOK Study
Brief Title: Assessment of the Impact of RNA Genomic Profile on Treatment Decision-making in HER2 Equivocal Breast Cancer Patients
Acronym: EQUIVOK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Take care recommendations for Her2 equivok patients has changed.
Sponsor: Centre Jean Perrin (Other)
Collaborators: Roche Pharma AG (Industry); NanoString Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A00240-53
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: Equivocal Her 2; Genomic test
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Cohort longitudinal follow up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of PAM 50 test in Her2 equivocal breast cancer patient (Experimental): Patients with an equivocal-HER2 breast cancer (IHC Score 2 and equivocal ISH defined as HER2/Chr17 ratio <2 and 4 ≤HER2 gene number copy < 6) will be eligible for RNA genomic test (PAM 50 test).
  Interventions: Diagnostic Test: PAM 50 test

INTERVENTIONS:
Diagnostic Test: PAM 50 test — Patients with an equivocal-HER2 breast cancer (IHC Score 2 and equivocal ISH defined as HER2/Chr17 ratio <2 and 4 ≤HER2 gene number copy < 6) will be eligible for RNA genomic test (PAM 50 test). The use of genomic test could help the oncologist to define the better therapeutic decision in a HER2 equivocal population.

SUMMARY:
The American Society of Clinical Oncology (ASCO) and the /College of American Pathologists (CAP) recommend that HER2 status (negative or positive) must be determined in all patients with invasive breast cancer. The knowledge of HER2 status will help the oncologist in prescribing or not a HER2-targeted therapy to patients. Presently, two main methods are used to assess HER2 status: immunohistochemistry (IHC, protein expression) and in situ hybridization (ISH, gene expression) in order to classify tumor sample as positive, negative or equivocal. When a tumor is classified HER 2+ by IHC method, a second test is performed using ISH methods (FISH, SISH, CISH). In case of HER2 equivocal result with ISH method (4 ≤HER2 gene number copy <6), the patient is eligible to an anti-HER2 therapy after discussed during MD-MM. This decision should be individualized on the basis of patient status (comorbidities and prognosis) and patient preferences after discussing available clinical evidence.

Based on molecular classification, RNA expression could help to discriminate breast cancer subtypes (luminal A, luminal B, HER2-overexpressed and triple negative). Prosigna is a genomic test, developed by NanoString® based on the PAM50 gene signature, which measures the expression of 50 genes to classify tumors into 1 of 4 intrinsic subtypes and could allow determining the HER2 status.

This study was designed in order to define if such a test could help the oncologist to define the better therapeutic decision in a HER2 equivocal population. In addition, concordance tests will be performed. The aim of this study is to assess the modification decision rate between the first and the second multidisciplinary decision-making meeting in HER2 equivocal patients using genomic testing.

ELIGIBILITY:
Inclusion Criteria:

* Performance status ≤ 2 (according to WHO criteria)
* Patient with early invasive breast cancer histologically confirmed stage I to IIIA)
* Positive or negative lymph node involvement
* Positive or negative Hormonal Receptors (Estrogens and/or Progesterone),
* Equivocal HER2 status (IHC Score 2 and equivocal ISH defined as HER2/Chr17 ratio <2 and 4 ≤ HER2 gene number copy < 6) as assessed on surgical specimen
* Adequate Hematological, Hepatic, Renal and Cardiac Functions
* Patient potentially eligible for an anti-HER2 therapy
* Patient eligible to receive an adjuvant therapy
* Signed Informed Consent
* Patient with social insurance.

Exclusion Criteria:

* Non-measurable tumor
* Unknown Hormonal Receptors
* Unknown node involvement
* Positive or negative HER2 status (Score 0, 1 or 3 IHC, or Negative or positive ISH)
* Disease stage ≥IIIB
* Patient not able to follow the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
The modification of therapeutical decision between the first and the second multidisciplinary decision-making meeting (MD-MM) using a genomic testing | The measure will be realised after the second multidisciplinary decision-making meeting that is about one month after patient's inclusion.
  Percentage of therapeutical strategy changes between the first and the second multidisciplinary decision-making meetings.

SECONDARY OUTCOMES:
The HER2 overexpression incidence according to RNA genomic profile among equivocal-HER2 patients | The measure will be done when the genomic test is realised, that is about three weeks after patient's inclusion.
  Percentage of HER2 classified patients using a genomic test among equivocal-HER2 patients
The concordance between the second multidisciplinary decision-making meeting decision and the HER2 genomic test result | The measure will be done when the genomic test is realised, that is about three weeks after patient's inclusion.
  Percentage of second multidisciplinary decision-making meeting decision in accordance with genomic test result and reasons justifying discrepancies (check-list and comments)

OTHER OUTCOMES:
To compare results from different ISH methods used | The measure will be done when the genomic test is realised, that is about three weeks after patient's inclusion..
  Comparison between all ISH (FISH, SISH, CISH, or DDISH) methods based upon the HER2-eligible classification (Wolff et al 2013)
The concordance between local and centralized anatomopathologist HER2 status | The measure will be done when the genomic test is realised,that is about three weeks after patient's inclusion.
  Concordance between local and centralized anatomopathologist HER2 status.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Ange MOURET-REYNIER, MD, Principal Investigator — Centre Jean Perrin
Locations (16):
- France (16):
  - CHRU Jean Minoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - CHU Albert Michalon, Grenoble
  - Hopital DUPUYTREN, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de Montpellier, Montpellier
  - Institut Jean Godinot, Reims
  - Institut du Cancer COURLANCY, Reims
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No